CLINICAL TRIAL: NCT07050888
Title: Effect of Inulin Supplementation on Glycaemic Control and Immunological Parameters in Type 1 Diabetes (2024)
Acronym: INCREASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Max Nieuwdorp, Principial investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024.1028
Record Dates: First submitted 2025-06-06; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; inulin; gut microbiome; prebiotics; CGM metrics; immunological parameters
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Inulin; Prebiotics

STUDY DESIGN:
Intervention Model Description: 2x38 participants will be randomly allocated to inulin or placebo once daily for 90 days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The unblinded researcher will provide the study intervention to the blinded investigator in a coded fashion. Both the investigator and the participant are blinded. In case of emergency, an unblinding protocol is activated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inulin (Experimental): prebiotic fermentable fiber inulin
  Interventions: Dietary Supplement: Inulin (prebiotic, fermentable fiber)
- Placebo (Placebo Comparator): Placebo: Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Inulin (prebiotic, fermentable fiber) — inulin (prebiotic, fermentable fiber)
  Arms: Inulin
Dietary Supplement: Placebo — placebo (matodextrin)
  Arms: Placebo

SUMMARY:
The goal is to establish the effect of oral inulin supplementation on continuous glucose monitoring (CGM) metrics and immunological parameters in adults with type 1 diabetes. The investigators will perform a double-blind, randomized, placebo-controlled trial in 2x38 participants to measure effects on CGM metrics, gut microbiome composition, residual beta cell and immunological parameters.

DETAILED DESCRIPTION:
The investigators perform a double-blind, randomized, placebo-controlled trial in 2x38 adults with type 1 diabetes. The participants will be given inulin or placebo once daily in powder, which can be dissolved in water and ingested orally, for 90 days. The main study endpoint is the difference in time in range between the groups between baseline and end-of-study. Secondary endpoints include changes in glycaemic variability, time in tight glycaemic range and hypoglycaemic episodes, gut microbiome composition, changes in residual beta cell function, changes in immunological parameters and validated questionnaires (Quality of Life and gastro-intestinal complaints).

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of type 1 diabetes, as made by their primary clinician
* A time in range of <80% in the last four weeks before screening

Exclusion Criteria:

* Use of any fibre supplementation (within the last month before screening or ongoing)
* Use of antibiotics in the lasts three months before screening or during study period
* Active infection during the study visit
* Inability or unwillingness to donate feces or urine.
* Illicit drug use (e.g. MDMA/amphetamine/cocaine/heroin/GHB) in the past three months or use during the study period.
* Inability or unwillingness to provide informed consent.
* Absence of a large bowel (ie colostomy)
* Active inflammatory bowel disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Time in range | 90 days
  Difference in time in range between the groups between baseline and end-of-study

SECONDARY OUTCOMES:
Continuous glucose monitoring | 90 days
  changes in glycaemic variability, time above range, time below range and hypoglycaemic episodes
Gut microbiome composition | 90 days
Residual beta cell function | 90 days
  Changes in urinary C-peptide-to-creatinine-ratio (UCPCR)
Immunological parameters | 90 days
  Plasma cytokines IFN-α, IFN-β, IFN-γ, IL-10 by ELISA
Gastrointestinal Symptom Rating Scale (GSRS) | 90 days
  Questionnaire. The minimum and maximum score are 15 and 105 points respectively, and a higher score in the scale reflects more gastro-intestinal complaints.
Dietary intake | 90 days
  Recorded of 3 days with "Eetmeter".
Gut inflammation | 90 days
  Fecal IgA and calprotectin in ug/g
CRP | 90 days
  C-reactive protein (mg/L)
Leukocyte (differentation) | 90 days
  ×10 9 /L
Diabetes autoantibodies anti-GAD, anti-IA2, anti-ZnT8 | 90 days
  units per milliliter (U/mL)
HbA1c | 90 days
  Millimoles of HbA1c per mole of hemoglobin (mmol/mol)
Quality of life questionnaire | 90 days
  Quality of life SF-12 v2 questionnaire, a higher score reflects higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nordin Hanssen, Principal Investigator, Principal Investigator — Amsterdam UMC
Locations (2):
- Netherlands (2):
  - Diabeter Centrum Amsterdam, Amsterdam
  - Amsterdam UMC, Amsterdam

IPD SHARING:
Plan to Share IPD: No